CLINICAL TRIAL: NCT01932684
Title: EFFECTS OF BREATH AND STACKING-SPIROMETRY INCENTIVE PACKAGES IN THE RIB CAGE IN PATIENTS WITH PARKINSON'S DISEASE
Brief Title: Effects Of Breath And Stacking-Spirometry Incentive in Patients With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Daniella Cunha Brandao, PhD, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Rhayssa dissertação
Record Dates: First submitted 2013-07-09; First posted 2013-08-30 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2012-12

CONDITIONS: Parkinson's Disease.
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Incentive spirometry (Experimental): Was utilized an incentive spirometer volume in this group.
  Interventions: Other: Incentive spirometry; Device: 5000 Voldyne ® Sherwood Medical, USA
- Control Group (No Intervention)
- Breath Stacking (Experimental): We used a face mask silicone connected to a check valve allowing only inspiration and is connected to a spirometer showed that the volume inspired by the individual.
  Interventions: Other: Breath-Stacking; Device: Silicone face mask

INTERVENTIONS:
Other: Breath-Stacking — We used a silicone face mask, connected to a unidirectional valve which allowed only inspiration and is connected to a spirometer showed that the volume inspired by the individual. The face mask was attached to the appraised performed successive breaths until the researcher realized the lack of volume of air being inhaled and this time it was allowed to expire (Baker et al., 1990; Feitosa et al., 2012).
  Arms: Breath Stacking
Other: Incentive spirometry — We used an incentive spirometer volume (5000 Voldyne ® Sherwood Medical, USA). Subjects performed slow, deep inhalations from functional residual capacity to total lung capacity, seeking to sustain the inspiration for at least three seconds (Restrepo et al., 2011).
  Arms: Incentive spirometry
Device: 5000 Voldyne ® Sherwood Medical, USA
  Arms: Incentive spirometry
Device: Silicone face mask
  Arms: Breath Stacking

SUMMARY:
Objective: To evaluate the effects of technical-Breath Stacking (BS) and incentive spirometry (IS) on the volume of the chest immediately after and within thirty minutes after the techniques in patients with Parkinson's disease (PD). Methods: This is a study of cross-over. The study investigated 14 patients with mild to moderate PD. The subjects performed the technique Breath-Stacking, incentive spirometry volume and participated in a phase control according to randomization. The volunteers were evaluated by opto-electronic plethysmography in four stages: before, immediately after fifteen and thirty minutes after the completion of the techniques. The investigators used a repeated measures ANOVA with post-hoc Tukey test for parametric variables, and the Friedman test with post-hoc Dunns for nonparametric variables. The level of significance was set at 5%, p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Regular pharmacological treatment with levodopa and / or medications antiparkinsonian.

Exclusion Criteria:

* Patients who had previous lung disease;
* Altered mental status indicated by the MMSE (Mini Mental State Examination;
* A change in medication during the study;
* Demonstrated inability to perform satisfactorily any of the collection procedures of the study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-06; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The variation of the total volume and compartmental between technique Breath-Stacking in patients with Parkinson's disease | 25 days
The variation of the total volume and compartmental in the technique incentive spirometry in patients with Parkinson's disease | 25 days

SECONDARY OUTCOMES:
The duration of the effects of technical-Breath Stacking and incentive spirometry in patients with Parkinson's disease | 25 days

CONTACTS AND LOCATIONS:
Overall Officials: RHAYSSA RH RIBEIRO, Msc, Principal Investigator — Universidade Federal do Rio Grande do Norte
Locations (2):
- Brazil (2):
  - Universidade Federal de Pernambuco, Recife, Pernambuco
  - Departamento de Fisioterapia-Universidade Federal de pernambuco, Recife, Pernambuco

REFERENCES:
- [Result] Baker WL, Lamb VJ, Marini JJ. Breath-stacking increases the depth and duration of chest expansion by incentive spirometry. Am Rev Respir Dis. 1990 Feb;141(2):343-6. doi: 10.1164/ajrccm/141.2.343. PMID 2301851
- [Result] Cala SJ, Kenyon CM, Ferrigno G, Carnevali P, Aliverti A, Pedotti A, Macklem PT, Rochester DF. Chest wall and lung volume estimation by optical reflectance motion analysis. J Appl Physiol (1985). 1996 Dec;81(6):2680-9. doi: 10.1152/jappl.1996.81.6.2680. PMID 9018522
- [Result] De Pandis MF, Starace A, Stefanelli F, Marruzzo P, Meoli I, De Simone G, Prati R, Stocchi F. Modification of respiratory function parameters in patients with severe Parkinson's disease. Neurol Sci. 2002 Sep;23 Suppl 2:S69-70. doi: 10.1007/s100720200074. PMID 12548348